CLINICAL TRIAL: NCT05840432
Title: Description of the Performance of a New Index for Hypotension Prediction During the Immediate Postoperative Period of Cardiac Surgery in the Intensive Care Unit
Brief Title: Hypotension Prediction During Cardiac Surgery Postoperative Period
Acronym: HPI-CCV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: PIC146-22_FJD
Record Dates: First submitted 2023-02-22; First posted 2023-05-03 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Hypotension
Keywords: hypotension prediction index; cardiac surgery; postoperative period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cardiac Surgery Postoperative Patients: Cardiac Surgery Postoperative Patients who are admitted to the intensive care unit after the surgery, from the surgical room
  Interventions: Device: Postoperative hypotension prediction index

INTERVENTIONS:
Device: Postoperative hypotension prediction index — Performance of the hypotension prediction index (HPI) in predicting hypotension episodes in the first 12 h of cardiac surgery postoperative

SUMMARY:
The goal of this observational study is to learn about the performance of a new index for hypotension prediction during the immediate postoperative period of cardiac surgery patients in the intensive care unit. The main questions it aims to answer are:

1. Is this new index, Hypotension Prediction Index, able to predict hypotension during the immediate postoperative period in cardiac surgery patients in the intensive care unit?
2. How frequent hypotension is during the immediate postoperative period of cardiac surgery patients in the intensive care unit? Participants will not receive any treatment beyond the usual clinical practice during the study. All patients will have an invasive arterial line that is part of the usual clinical practice. This arterial line is connected to a pressure transducer for continuous measurement of arterial pressure. A transducer equipped with the necessary technology to calculate the hypotension prediction index will be used instead of the usual transducer. An echocardiogram will be performed in every patient in the study. This test is done frequently in patients after a cardiac surgery.

DETAILED DESCRIPTION:
A non-interventional study will be performed, in which physiological signals will be acquired using usual clinical practice monitoring devices. These devices will be connected to catheters that are used as a routine management of the study patients. No management indication will be performed as part of the study.

The patients who accepted to participate in the study by previously signing the informed consent, will be received at the intensive care unit coming from the surgical room after a programmed cardiac surgery and once stability is ensured, investigators will proceed to connect an arterial pressure catheter that is routinely inserted into the radial artery to an Acumen IQ sensor (Edwards Lifesciences, Irvine California, USA). This sensor replaces the pressure transducer normally used in clinical practice, has similar characteristics and its use does not interfere with the usual routine. This sensor will be connected to the multiparametric monitor situated at the patient's bedside and to the Hemosphere monitoring platform (Edwards Lifesciences, Irvine California, USA). Besides being used as a pressure transducer, the Acumen IQ sensor allows for a more detailed arterial pressure signal analysis together with the Acumen Hypotension Prediction Index software. This software automatically calculates every 20 seconds the HPI, the main study parameter of this project, which as previously mentioned predicts hypotension episodes (defining hypotension as mean arterial blood pressure below 65 mmHg for at least 1 minute). Besides the HPI, the Acumen Hypotension Prediction Index software calculates complementary hemodynamic monitoring parameters that can help managing patients with different conditions among which there an be found the moderate and high risk postoperative conditions. These parameters are: stroke volume, stroke volume variation, mean arterial pressure, dP/dt (the maximal of the first derivative during the ascending phase of the arterial pressure - time curve, related to the left ventricular contractility), cardiac index, systemic vascular resistance and arterial dynamic elastance (the ratio between the pulse pressure variation and the stroke volume variation, which allows to evaluate the afterload).

The study time will be 12 hours (counting from the moment of the beginning of the patient monitoring in the intensive care unit), during which, besides the parameters calculated by the Acumen Hypotension Prediction Index, monitoring clinical and analytical routine parameters will be collected as furtherly detailed. Moreover, a transthoracic echocardiogram will be routinely performed during the first 6 hours of the patient's stay in the intensive care unit. This is a noninvasive procedure and will not interfere with the patient's usual care.

The HPI will not be shown on the monitoring platform to avoid any influence on the normal clinical practice and to be able to measure the real incidence of hypotension episodes. The complementary parameters calculated by the software will be available to the treating physician and can be used for decision making based on his criteria. The results of the echocardiogram will be available as well to the treating physician and will be interpreted and used based on treating physician criteria.

As described, besides the evaluation of the HPI performance, the results of this study will allow to have information regarding the behavior of arterial pressure in cardiac surgery postoperative patients and the creation of a protocol to reduce hypotension in these patients.

Variables

The following variables will be studied:

* Epidemiologic: age, sex, weight, height.
* Severity and risk assessment and classification systems: APACHE II, EUROSCORE II, Sequential Organ Failure Assessment Score (SOFA), Simplified Acute Physiology Score III (SAPS III)
* Risk factors: renal failure, hypertension, diabetes, dyslipidemia
* Surgery: type, total surgery time, circulatory bypass time, ischemia time
* Monitoring: HPI, arterial pressure (mean, systolic, diastolic), stroke volume variation, pulse pressure variation, dynamic arterial elastance, dP/dt, cardiac index, central venous pressure, at admission and 12h later, besides variability analysis of these parameters. Continuous arterial pressure register will be analyzed and mean arterial pressure below 65 mmHg will be determined, normalized by the monitoring time.
* Hypotension treatment: fluid bolus, vasoactive and inotropic types and doses. This management will be performed according to physician criteria.
* Echocardiographic variables: right ventricle (RV) diameter /left ventricle (LV) diameter, Tricuspid Annular Plane Systolic Excursion (TAPSE), S wave, RV/LV ratio, pulmonary artery systolic pressure (PASP) estimation, LV ejection fraction, Left Ventricular Outflow Tract Velocity Time Integral (LVOT VTI), Right Ventricular Outflow Tract Velocity Time Integral (RVOT VTI), Pulmonary Velocity Acceleration Time (PVAT), inferior vena cava (IVC) diameter.
* Mechanical ventilation at admission and 12h later: positive end expiratory pressure (PEEP), FiO2 - Fraction of inspired oxygen (FiO2), tidal volume (VT), respiratory rate, mean pressure, plateau pressure, peak pressure.
* Blood analysis: hemoglobin, leukocytes, lymphocytes, arterial blood gas parameters, renal function, ferritin, D-dimer, interleukin 6 (IL-6), peak creatin kinase (CK), creatin kinase myocardial band (CK-MB), troponin I, brain natriuretic peptide (BNP).
* Clinical results: ICU length of stay, hospital length of stay, mechanical ventilation time, vasoactive support, and mechanical ventilation. Acute kidney failure development, peak troponin I, perioperative acute myocardial infarction, mortality, stroke, evolutive SOFA, other complications (sepsis)

Data Analysis

The adequate analytic and statistical methods will be used to:

* Describe arterial pressure and complementary hemodynamic variables behavior
* Evaluate HPI performance predicting hypotension in the postoperative cardiac surgery period in the intensive care unit
* Create a predictive model for hypotension development in the cardiac surgery postoperative period
* Analyze the relationship between postoperative hypotension and complications development.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 y.o.
* Programmed cardiac surgery
* Hemosphere platform availability
* Signed informed consent

Exclusion Criteria:

* Need for circulatory or respiratory mechanical assistance device support
* Urgent/emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients in the postoperative period of programmed cardiac surgery, who are admitted to the intensive care unit after the surgery. according to inverstigator and Hemosphere monitor disponibilty
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
HPI Performance on Hypotension Prediction | First 12 hours of the cardiac surgery postoperative period
  Area Under the Receiver Operator Characteristic (ROC) curve for hypotension prediction, defining hypotension as mean arterial blood pressure below 65 mmHg for at least 1 minute.

SECONDARY OUTCOMES:
Hypotension incidence | First 12 hours of the cardiac surgery postoperative period
  Hypotension incidence
Hypotension consequences: acute kidney injury | Up to two months after surgery
  Development of Acute kidney injury described as an increase in Serum Creatinine (SCr) by ⩾0.3 mg/dl (⩾26.5 μmol/l) within 48 hours or Increase in SCr to ⩾1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or Urine volume <0.5 ml/kg/h for 6 hours, as well as maximum creatinine levels.
Hypotension consequences: myocardial injury | First 7 days of ICU admission
  Development of complications related with hypotension such as myocardial injury. Dynamics of Troponin I levels will be studied, baseline at ICU admission, peak levels, dynamics during the first 12h hours of admission up to the first 7 days of ICU admission.
Hypotension consequences: prolonged mechanical ventilation | Mechanical ventilation free days at 2 months
  Development of complications related with hypotension such as prolonged mechanical ventilation defined as more than 21 days of mechanical ventilation.
Actions performed for hypotension management: vasopressors and inotropic drugs | First 12 hours of the cardiac surgery postoperative period
  Administration of noradrenaline, dobutamine, levosimendan and vasopressin accumulated dosis and maximum dosis
Actions performed for hypotension management: fluid therapy | First 12 hours of the cardiac surgery postoperative period
  Description and quantification of actions performed for hypotension management such fluid therapy type and dose in ml/h.
General outcomes: Intensive care unit and hospital length of stay | Up tp two months after surgery
  The intensive care unit length of stay (days) and hospital length of stay (days) will be studied
General outcomes: mortality | Up to two months after surgery
  Mortality (binary variable, alive or dead) will be studied
General outcomes: respiratory failure | Up to two months after surgery
  Respiratory failure development will be studied defined as failure to wean from mechanical ventilation within 48 hours of surgery or unplanned intubation/reintubation postoperatively.
General outcomes: nosocomial infections | Up to two months after surgery
  Nosocomial infections development will be studied, defined as an infection acquired during the process of receiving health care that was not present during the time of admission.
General outcomes: reintervention | First 48 hours of the cardiac surgery postoperative period
  Need for cardiac surgery reintervention (binary variable)

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit. Hospital Universitario Fundación Jimenez Diaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
In this study exists a potential generation of intellectual property generation.

REFERENCES:
- [Background] Guarracino F, Habicher M, Treskatsch S, Sander M, Szekely A, Paternoster G, Salvi L, Lysenko L, Gaudard P, Giannakopoulos P, Kilger E, Rompola A, Haberle H, Knotzer J, Schirmer U, Fellahi JL, Hajjar LA, Kettner S, Groesdonk HV, Heringlake M. Vasopressor Therapy in Cardiac Surgery-An Experts' Consensus Statement. J Cardiothorac Vasc Anesth. 2021 Apr;35(4):1018-1029. doi: 10.1053/j.jvca.2020.11.032. Epub 2020 Nov 19. PMID 33334651
- [Background] Fischer GW, Levin MA. Vasoplegia during cardiac surgery: current concepts and management. Semin Thorac Cardiovasc Surg. 2010 Summer;22(2):140-4. doi: 10.1053/j.semtcvs.2010.09.007. PMID 21092891
- [Background] Levin MA, Lin HM, Castillo JG, Adams DH, Reich DL, Fischer GW. Early on-cardiopulmonary bypass hypotension and other factors associated with vasoplegic syndrome. Circulation. 2009 Oct 27;120(17):1664-71. doi: 10.1161/CIRCULATIONAHA.108.814533. Epub 2009 Oct 12. PMID 19822810
- [Background] Ouattara A, Boccara G, Kockler U, Lecomte P, Leprince P, Leger P, Riou B, Rama A, Coriat P. Remifentanil induces systemic arterial vasodilation in humans with a total artificial heart. Anesthesiology. 2004 Mar;100(3):602-7. doi: 10.1097/00000542-200403000-00021. PMID 15108975
- [Background] Kotani Y, Yoshida T, Kumasawa J, Kamei J, Taguchi A, Kido K, Yamaguchi N, Kariya T, Nakasone M, Mikami N, Koga T, Nakayama I, Shibata M, Yoshida T, Nashiki H, Karatsu S, Nogi K, Tokuhira N, Izawa J. The impact of relative hypotension on acute kidney injury progression after cardiac surgery: a multicenter retrospective cohort study. Ann Intensive Care. 2021 Dec 20;11(1):178. doi: 10.1186/s13613-021-00969-4. PMID 34928430
- [Background] de la Hoz MA, Rangasamy V, Bastos AB, Xu X, Novack V, Saugel B, Subramaniam B. Intraoperative Hypotension and Acute Kidney Injury, Stroke, and Mortality during and outside Cardiopulmonary Bypass: A Retrospective Observational Cohort Study. Anesthesiology. 2022 Jun 1;136(6):927-939. doi: 10.1097/ALN.0000000000004175. PMID 35188970
- [Background] Weis F, Kilger E, Beiras-Fernandez A, Nassau K, Reuter D, Goetz A, Lamm P, Reindl L, Briegel J. Association between vasopressor dependence and early outcome in patients after cardiac surgery. Anaesthesia. 2006 Oct;61(10):938-42. doi: 10.1111/j.1365-2044.2006.04779.x. PMID 16978306
- [Background] Parke RL, McGuinness SP, Gilder E, McCarthy LW. Intravenous fluid use after cardiac surgery: a multicentre, prospective, observational study. Crit Care Resusc. 2014 Sep;16(3):164-9. PMID 25161017
- [Background] Meng L, Yu W, Wang T, Zhang L, Heerdt PM, Gelb AW. Blood Pressure Targets in Perioperative Care. Hypertension. 2018 Oct;72(4):806-817. doi: 10.1161/HYPERTENSIONAHA.118.11688. No abstract available. PMID 30354725
- [Background] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Background] Davies SJ, Vistisen ST, Jian Z, Hatib F, Scheeren TWL. Ability of an Arterial Waveform Analysis-Derived Hypotension Prediction Index to Predict Future Hypotensive Events in Surgical Patients. Anesth Analg. 2020 Feb;130(2):352-359. doi: 10.1213/ANE.0000000000004121. PMID 30896602
- [Background] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827